CLINICAL TRIAL: NCT03245489
Title: Pembrolizumab in Combination With Anti-platelet Therapy for Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Anti-platelet + Pembro for H&N Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 102727
Record Dates: First submitted 2017-06-13; First posted 2017-08-10 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — pembrolizumab; Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Group 1 will be treated with Regimen A, followed by Regimen B. Regimen A is pembrolizumab, ASA and clopidogrel daily for 6 weeks. Regimen B is pembrolizumab alone for 6 weeks.
  Interventions: Drug: Pembrolizumab; Drug: Clopidogrel; Drug: acetylsalicylic acid
- Group 2 (Experimental): Group 2 will be treated with Regimen B, followed by Regimen A. Regimen B is pembrolizumab alone for 6 weeks. Regimen A is pembrolizumab, ASA and clopidogrel daily for 6 weeks.
  Interventions: Drug: Pembrolizumab; Drug: Clopidogrel; Drug: acetylsalicylic acid

INTERVENTIONS:
Drug: Pembrolizumab — 200mg intravenous (IV) over 30 minutes
  Other Names: Keytruda
Drug: Clopidogrel — 75mg/day oral
  Other Names: Plavix
Drug: acetylsalicylic acid — 81mg/day oral
  Other Names: ASA; aspirin

SUMMARY:
The purpose of this study is to see if anti-platelet therapy combined with anti-PD-1 immunotherapy can cause a more favorable immunologic response thatn with immunotherapy alone in patients with recurrent or metastatic squamous cell carcinoma of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has pathologic confirmation of recurrent or metastatic HNSCC, regardless of HPV status.
2. Subject has tumor that expresses PD-L1 (Combined Positive Score [CPS] > 1) as determined by an FDA-approved test or subject has experienced disease progression on or after platinum-containing chemotherapy.
3. Subject's scans have been reviewed at head and neck tumor board to assess tumor involvement.
4. Subject is 18 years of age or older.
5. Subject has measurable disease according to RECIST 1.1. Tumor lesions situated in previously irradiated areas are considered measurable if progression has been demonstrated in such lesions.
6. Subject has an ECOG performance status of 0 to 2
7. Subject has estimated life expectancy of at least 3 months.
8. Subject has adequate hematologic function, defined as:

   1. ANC >1000 K/CUMM
   2. Hemoglobin >8.0 Grams/dL
   3. Platelets >75,000 K/CUMM
   4. INR < 1.7
9. Subject has adequate renal function, defined as estimated creatinine clearance > 30 mL/min according to the Cockcroft-Gault formula.
10. Subject has adequate hepatic function, defined as:

    1. Total bilirubin ≤ 1.5 x ULN
    2. AST and ALT ≤ 2.5 x ULN
11. Female and male subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication. Effective forms of contraception include abstinence, hormonal contraceptive in conjunction with a barrier method, or a double barrier method. Women of non-child-bearing potential may be included if they are either surgically sterile or have been post-menopausal for > 1 year.

Note: Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 14 days of registration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Exclusion Criteria:

1. Subject is receiving concomitant immunosuppressive therapy, defined as:

   1. Immunosuppressants, including: tacrolimus, sirolimus, everolimus, cyclosporine, azathioprine, mycophenolate mofetil, antithymocyte globulin, basiliximab, belatacept
   2. Systemic corticosteroids (except for short term treatment of allergic reactions or for treatment of irAE). Steroids with no or minimal systemic effect (topical, inhalation) are allowed.
   3. Chemotherapy
   4. Immunotherapy
   5. Monoclonal antibodies
2. Concurrent anticancer treatment within 14 days before the start of trial treatment.
3. Subject has had major surgery within the last 28 days.
4. Subject has an underlying bleeding disorder.
5. Subjects requiring re-irradiation to head and neck.
6. Subject is receiving anticoagulation (see section 7.2 for medication examples). Subjects must have a washout period of 7 days from registration.
7. Subject has HNSCC with abutment or encasement of the internal carotid artery, external carotid artery or common carotid artery or any of the arterial branches.
8. Subject has a draining fistula or wound in the head/neck.
9. Subject with known aneurysm or pseudoaneurysm of the head/neck related to surgery.
10. Subject has uncontrolled CNS metastases. Subjects with previously treated brain metastases will be allowed if the brain metastases have been stable without CNS-directed therapy (such as radiation or surgery) or steroid treatment for for at least 4 weeks prior to registration.
11. Receipt of any organ transplantation.
12. Active or history of any autoimmune disease (except type I DM, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment, which are allowed) or immunodeficiencies.
13. Known severe hypersensitivity reactions to monoclonal antibodies (grade ≥ 3NCI-CTCAE v4.0), any history of anaphylaxis or uncontrolled asthma.
14. Subjects who have a hypersensitivity to aspirin or NSAIDs.
15. Concurrent NSAID therapy (see section 7 for examples). Subjects must have a washout period of 7 days from registration.
16. Subjects with an acute gastrointestinal ulcer.
17. Subjects with active hemorrhagic diathesis.
18. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (NYHA class ≥ II), or serious uncontrolled cardiac arrhythmia.
19. All other significant diseases, which in the opinion of the investigator, may impair the subject's tolerance of trial treatment.
20. Vaccination within 4 weeks of the 1st dose of pembrolizumab and while on study is prohibited EXCEPT for administration of inactivated vaccines (e.g. inactivated influenza vaccine).
21. Women who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Effect of Pembro + antiplatelet on major cellular parameters | 12 weeks
  Immunologic response profile will be measured by changes in major cellular parameters in peripheral blood mononuclear cells pheotyped by flow cytometry for MDSCs, T and B cell activation markers and polyclonal IFNy-production by CD4 and CD8 response after P/I stimulation) in pembrolizumab alone and pembrolizumab + antiplatelet therapy. Markers will be measured at baseline, end of the first regimen and end of the second regimen. Changes in cellular parameters from the previous timepoint will be evaluated using a repeated measures ANOVA model. Cellular parameters will be evaluated in aggregate to report the immunologic response.

SECONDARY OUTCOMES:
Effect of Pembro + antiplatelets on immunologic markers | 12 weeks
  Immunologic markers will be measured in patients who have been treated with two cycles of pembrolizumab alone and who are pembrolizumab naive. Markers will be evaluated by looking at phyenotyping by flow cytometry and changes of 65-panel systemic cytokines and chemokine levels. Markers will be measured at baseline, end of the first regimen and end of the second regimen. Changes to markers will be reported in aggregate to show the overall immunologic effect of the combination of pembrolizumab + Anti-platelets in patients.
Frequency of adverse events reported | 12 weeks
  Safety data will be tabulated by type and grade of adverse event and will use CTCAE v. 4.0
Tumor response rate | 12 weeks
  Objective response will be evaluated with computed tomography (CT) of the neck, chest and abdomen at baseline and post-treatment using RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: John Kaczmar, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No